CLINICAL TRIAL: NCT04134390
Title: Pilot Study of Cabozantinib Efficacy, Safety and Tolerability in Metastatic Renal Carcinoma in Aged Fragile Patients: CABOMAYOR Study
Brief Title: Study of Cabozantinib Efficacy, Safety and Tolerability in Metastatic Renal Carcinoma in Aged Fragile Patients: CABOMAYOR Study
Acronym: CABOMAYOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABOMAYOR; 2019-001639-30 (EudraCT Number)
Record Dates: First submitted 2019-10-15; First posted 2019-10-22 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Old Age; Debility; Renal Carcinoma Metastatic
Keywords: fragile; renal carcinoma; old age
MeSH Terms: conditions — Frailty; Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Cabozantinib 40 mg per os (p.o.) once daily in 28-day cycles. Dose can be escalated to 60 mg to avoid suboptimal exposure to the drug if 40 mg is considered tolerated. If the dose of 40 mg is not tolerated, a de-escalation to 20 mg, temporary interruption, or stopping cabozantinib will be possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Cabozantinib 40 mg p.o. once daily in 28-day cycles.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Subjects will receive cabozantinib 40mg p.o. as long as they continue to experience clinical benefit or until unacceptable toxicity, the need for alternative anticancer treatment, or other reasons for treatment discontinuation

SUMMARY:
Aged fragile patients are not usually included in clinical trials and efficacy and tolerability of the different available treatments in this population are unknown.

Conversely, ageing has been associated with a decrease in the efficacy of immune checkpoint inhibitors due to a decline in the effectiveness of the immune system (immunosenescence). In the Checkmate 025 trial comparing nivolumab with everolimus, the Hazard Ratio (HR) in patients older than 75 years old favoured everolimus, 1.23 (0.66-2.31). Thus, TKis might be a better treatment option for this population. However, the absence of data and concerns about possible secondary effects associated, can preclude clinicians to treat aged fragile patients with cabozantinib. A pilot phase II trial would help to have data on safety and efficacy of cabozantinib in this aged fragile population.

In METEOR trial around 60% of patients reduced the dose of cabozantinib because of toxicity and tolerance problems. It is suspected that the efficacy of cabozantinib in the population to be included in this trial (aged and fragile) will be similar to that observed in CABOSUN trial (disease control rate around 75%). However, there is no information available in this group of patients. On the other hand, in the >75 years old subgroup within the METEOR trial, 37% discontinued due to adverse events, 85% needed dose reductions and median average daily dose was 33,6 mg. For this reason, the cabozantinib initial dose chosen for patients to be included in this study is 40 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. Documented histological or cytological diagnosis of renal cell cancer.
2. Measurable disease per RECIST 1.1 as determined by the investigator.
3. Metastatic disease.
4. Patient must have signed the informed consent document.
5. Capable of understanding and complying with the protocol requirements.
6. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) 0-2.
7. Patients aged >70 years old with Society of Geriatric Oncology (SIOG) defined fragile population or patients >75 years with or without SIOG defined fragility.
8. No previous treatment for Metastatic Renal Cell Carcinoma (mRCC)
9. Adequate organ function based on standard laboratory tests including haematology, serum chemistry, lipids, coagulation, thyroid function, and urinalysis.
10. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.

Exclusion Criteria:

1. Previous treatment for mRCC.
2. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before inclusion.
3. Known brain metastases or cranial epidural disease unless adequately treated and stable for at least 3 months before inclusion.
4. Concomitant anticoagulation at therapeutic doses with oral anticoagulants or platelet inhibitors or low molecular weight heparins (LMWH).
5. Chronic treatment with corticosteroids or other immunosuppressive agents
6. Uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions: Cardiovascular disorders, Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation, Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 3 months before inclusion, Cavitating pulmonary lesion(s) or known endobronchial disease manifestation and/or Lesions invading major pulmonary blood vessels.
7. Major surgery within 2 months before inclusion.
8. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 msec within 10 days before inclusion.
9. Inability to swallow tablets or capsules.
10. Previously identified allergy or hypersensitivity to components of the study treatment formulation.
11. Diagnosis of another malignancy within 2 years before inclusion, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  Complete Response (CR) evaluated by Evaluation Criteria In Solid Tumors (RECIST) 1.1 according to investigator criteria.
Objective Response Rate (ORR) | Up to 24 months
  Partial Response (PR) evaluated by Evaluation Criteria In Solid Tumors (RECIST) 1.1 according to investigator criteria.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 24 months
  Adverse Events (AEs) experienced by patients. AEs will be assessed according to National Cancer Institute-Common Terminology Criteria (NCI-CTC) v 5.0 criteria.
Disease Control Rate (DCR) | Up to 24 months
  Complete Response (CR) evaluated by RECIST 1.1 criteria according to investigator criteria.
Disease Control Rate (DCR) | Up to 24 months
  Partial Response (PR) evaluated by RECIST 1.1 criteria according to investigator criteria.
Disease Control Rate (DCR) | Up to 24 months
  Stable Disease (SD) evaluated by RECIST 1.1 criteria according to investigator criteria.
Progression Free Survival (PFS) | Since the patient's study enrolment until patient progression, assessed up to 24 months
  Time in months since the patient's study enrolment until patient progression according to RECIST 1.1 criteria
Overall Survival (OS) | Since the patient's study enrolment until death assessed up to 24 months
  It is time in months since the patient's study enrolment until death

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Climent, MD, Principal Investigator — FIVO
Locations (10):
- Spain (10):
  - Hospital de Ciudad Real, Ciudad Real
  - ICO L'Hospitalet, L'Hospitalet de Llobregat
  - Hospital Insular de Gran Canarias, Las Palmas de Gran Canaria
  - Hospital Lucus Augusti, Lugo
  - Hospital Infanta Sofia, Madrid
  - Hospital Universitario de Donostia, San Sebastián
  - Fundación Instituto Valenciano de Oncologia, Valencia
  - Hospital Doctor Peset, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided